CLINICAL TRIAL: NCT01425437
Title: Keloid Tissue Bank - Longitudinal Clinical Data Repository; A Genomic and Molecular Research to Identifying Molecular Markers and Signal Transduction Pathways in Keloid; and Correlations With the Natural History of the Disease.
Brief Title: Keloid Tissue Bank
Status: Terminated | Type: Observational
Why Stopped: Poor Enrollment
Sponsor: Tirgan, Michael H., M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: Tirgan 11-02
Record Dates: First submitted 2011-08-23; First posted 2011-08-30 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Keloid
Keywords: Keloid
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sample of keloid tissue and small amount of normal appearing skin from an area that is adjacent to the keloid will be collected from each participant. Each patient may undergo one or more biopsies during the span of this study. Tissue biopsy may be repeated from the same or a different keloid in the same patient. Patients may be re-contacted for additional blood or other tissue samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with keloid: All patients will have a clinical diagnosis of keloid and will consent to participate in this study.

SUMMARY:
Much progress in treatment of various tumors has been made in the laboratory and the results have been brought back to the patients, i.e. from bench to bedside. This trial intends to collect samples of keloid tissue from patients and study them in laboratory. Such a research may help us with finding better treatments for keloid.

DETAILED DESCRIPTION:
To aims of this trial are:

1. To prospectively collect keloid and normal skin tissue samples from patients with keloid by performing keloid tissue biopsy and biopsy of uninvolved skin.
2. To collect blood and/or saliva for genomics, proteomics, tissue culture, flow cytometery and other keloid investigational studies.
3. To collect any keloid tissue that has been previously removed from the patient (unrelated to enrollment on this study).
4. To prospectively collect keloid tissue from patients who are undergoing a planned surgical removal of their keloids.
5. To evaluate keloid histology, genomics, proteomics, molecular markers, cytokines, growth factors receptors, ligands and signal transduction pathways within keloid tissue in order to find druggable targets.
6. To prospectively follow the patients and correlate patient demographics and natural history of the disease, response to the past and future treatments with the genomic and molecular maker profiles.
7. To culture nucleated blood cells from keloid patients in order to determine the genomics of this disease as well as learning about potential presence of keloid stem cell in peripheral blood. To use flow cytometry as well as other technology to search for circulating keloid stem cells in peripheral blood.
8. To test in vitro:

A- The effect of small molecule kinase inhibitors on the activation of wild-type and mutant kinases.

B- The effects of various drugs that inhibit ligands, receptors or pathways.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have clinically confirmed diagnosis of keloid
2. Signed consent form; parent or a legal guardian should consent for children and those under age of 18.
3. Have at least one paraffin block of excess keloid tissue that has been removed in the past; or is planned to be removed in future.
4. Able and willing to undergo a keloid biopsy (optional)
5. Able and willing to undergo biopsy of their normal appearing skin (optional, minimum age 18).

Exclusion Criteria:

1. Individuals who are mentally challenged, who cannot consent to participate in this study.
2. Psychological Illness that may result in non-compliance with the procedure and the required follow up.
3. Known allergy to lidocaine or other local anesthetics.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with a clinical diagnosis of keloid who are 13 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2012-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of cases with a genetic mutations within the study cohort will be measured. | Three years
  Prevalence of various biomarkers and/or mutations will be determined and co-related with the clinical presentation of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Tirgan, MD, Study Chair — Keloid Research Foundation
Locations (1):
- Michael H. Tirgan, MD, New York, New York, United States